CLINICAL TRIAL: NCT04300088
Title: A Prospective Study of the Relevance of the HLA-G Immune Checkpoint in Cancer Immunotherapy
Acronym: GEIA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190362
Record Dates: First submitted 2020-03-04; First posted 2020-03-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Solid Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with advanced solid cancer treated with anti-PD(L)1: Adult patients with advanced solid cancer treated with anti-PD(L)1 immunotherapy with or without anti-CTLA4 immunotherapy.

SUMMARY:
Therapeutic targeting of immune checkpoints PD-1/PD-L1 and/or CTLA-4 is efficient in several solid cancer subtypes, however only some patients do experience clinical benefit from these treatments. One explanation could be that multiple redundant checkpoints are present within the tumor, simultaneously keeping in check the patient's immune response. The immune checkpoint HLA-G is neo-expressed in over 50% of cases in some cancer subtypes and associated with more dismal prognosis. The immunosuppressive effects of HLA-G may result in resistance to current immunotherapy drugs.

The GEIA study explores the impact of HLA-G tumor expression on the efficacy of cancer immunotherapy in solid cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Social insurance
* Ability to provide signed consent
* Histologically proven solid cancer (non-small cell lung cancer, urothelial carcinoma, renal cell carcinoma, other)
* Advanced and/or metastatic disease not accessible to local treatment
* At least one target lesion according to iRECIST
* Available fixed tumor sample for immunohistochemistry studies
* Treatment with anti-PD(L)1 immunotherapy with or without anti-CTLA4 immunotherapy

Exclusion Criteria:

* Women pregnant or breastfeeding
* Inability to consent to this research
* Previous cancer immunotherapy (except BCG instillations for non-muscle infiltrative bladder cancer)
* Patients chronically infected with HIV, HBV or HCV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with advanced solid cancer treated with anti-PD(L)1 immunotherapy with or without anti-CTLA4 immunotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 281 (Estimated)
Dates: Start 2020-03-10 (Estimated); Primary Completion 2020-09-10 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Objective tumor response rate | at 6 months
  The impact of HLA-G tumor expression (evaluated by immunohistochemistry) on tumor response rates (evaluated with iRECIST) in solid cancer patients treated with anti-PD(L)1 immunotherapy with or without anti-CTLA4 immunotherapy.

SECONDARY OUTCOMES:
Progression free-survival | at 6 months
Progression free-survival | at 1 year
Progression free-survival | at 2 years
Overall survival | at 6 months
Overall survival | at 1 year
Overall survival | at 2 years
Specific disease survival | at 6 months
Specific disease survival | at 1 year
Specific disease survival | at 2 years
Incidence of adverse events | at 2 years
  Adverse events will be assessed using Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Soluble HLA-G levels counts | Up to 24 months
  Soluble HLA-G levels will be evaluated by ELISA.The correlation between tumor HLA-G expression and soluble HLA-G levels will be studied.

IPD SHARING:
Plan to Share IPD: Undecided